CLINICAL TRIAL: NCT02767908
Title: Randomised Controlled Trial to Test the Effectiveness of an Intensive Home Support Intervention for Newly Abstinent Smokers Leaving Hospital
Brief Title: Hospital to Home, Smoker Support Trial
Acronym: HTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16022; RP-PG-0608-10020 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2016-05-06; First posted 2016-05-11 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2017-08

CONDITIONS: Smoking Cessation
Keywords: Tobacco; Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Participants in the usual care group will be offered and, if accepted, provided with smoking cessation support that meets the recommendations of NICE PH48 guidance including pharmacotherapy and behavioural support before leaving hospital, referral to NHS SSS for continued care after discharge, and ascertainment of smoking status at 4 weeks; participants will also be asked to consent to smoking status ascertainment at three months. Those who report cessation at 4 weeks and/or three months will be requested to agree to a home visit for CO validation. All will be asked at four weeks and 3 months to list the cessation support, in terms of pharmacotherapy and behavioural support from local or other services, delivered since the last contact.
- Intervention (Active Comparator): A home visit will be carried out as soon as practicable after discharge and typically within 48 hours, to deliver a multi-component intervention. Intervention components all have an existing evidence base proving or suggesting potential efficacy for smoking cessation and/or relapse prevention, though their feasibility and importance when delivered as a combined package have not been tested.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Participants will receive a tailored support package which will include; Nicotine replacement products, behavioural support, including telephone support, Carbon dioxide measurements, home air quality measurements, signposting to support groups, and self-help materials.For participants who decline a home visit, the above support options will be offered as far as possible through telephone contact and delivered to the extent accepted by the participant. Those who report cessation at 4 weeks and/or three months will be requested to agree to a home visit for CO validation.
  Arms: Intervention

SUMMARY:
The present study is proposed to build on the investigators demonstration of the effectiveness of default delivery of smoking interventions in hospital inpatients by testing a multi-component intervention to prevent relapse to smoking after hospital discharge. The proposed intervention is designed to integrate easily with existing services, and hence be widely implemented if shown to be effective

DETAILED DESCRIPTION:
The Investigators analysis of electronic primary care records has recently estimated that approximately 1.1 million smokers are admitted to English hospitals every year . Every one of these admissions represents a prime opportunity to intervene to promote smoking cessation, particularly since most smokers abstain from smoking while in hospital. Recent NICE guidance (PH48) recommends that smoking cessation interventions should be provided in routine care pathways for all smokers admitted to hospital; The Investigators earlier work (Evaluation of the impact of a systematic delivery of cessation interventions on delivery of smoking cessation in secondary care. REC Reference Number:10/H0403/34) in this Programme (RP-PG-0608-10020) has demonstrated that default delivery of cessation support to all smokers in hospital significantly increases uptake of support and doubles the proportion of smokers who quit long term. Clinical experience indicates that many smokers admitted to hospital, particularly those with an illness caused or exacerbated by smoking, are motivated not to smoke again after discharge but are also likely to be heavily dependent on smoking and in many cases are disabled by lung or heart disease, socially isolated, and socio-economically deprived. On leaving hospital, many participants returned to a home environment where smoking has been an integral part of daily life for many years. It is therefore not surprising that whilst many participants managed to stay smoke-free during their hospital stay, relapse after discharge is common.

The Investigators previous study, among smokers who received care similar to that now recommended by NICE, 62% of participants abstinent at discharge had relapsed by 4 weeks, and 81% by 6 months. The Investigators hypothesise that many of these relapses could be prevented by interventions that help to sustain cessation and the maintenance of smoke-free home after discharge.

The investigators therefore propose to test the effectiveness of an intensive home support intervention for newly-abstinent smokers leaving hospital and involving home visits to support cessation and establishment of a smoke-free home; ensure receipt and correct use of smoking cessation pharmacotherapy; deliver behavioural support or else, where local services are preferred, transfer to local community Stop Smoking Services (SSS).

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 and over (with no upper age limit).
* Have been admitted for 24 hours or more to any participating inpatient ward at Nottingham City Hospital.
* Who report that they are current smokers, or had smoked within 7 days before the current admission.
* Are capable of understanding and consenting to the trial.

Exclusion Criteria:

* • If they are pregnant; Pregnant smokers (of whom very few are admitted to medical wards) will be offered cessation advice in line with NICE PH48 guidance.

  * If they do not consent to participate,
  * If they are too ill or otherwise lack capacity to understand the information and consent forms.
  * If they live more than 50 miles from the City Hospital (these patients will be referred to their local community cessation services, in line with NICE recommendations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Self-reported continuous smoking cessation since discharge | 4 weeks
  At four weeks post-discharge, validated by exhaled CO less than 6ppm

SECONDARY OUTCOMES:
Self-reported continuous cessation at three months post-discharge, validated by exhaled CO less than 6ppm | 12
  At 12 weeks post-discharge, validated by exhaled CO less than 6ppm
Un-validated self-reported continuous smoking cessation at four weeks | 4 weeks
  Individual declares "No" to smoking any form of tobacco product since being discharged from hospital
Un-Validated Self-reported continuous cessation at three months post-discharge | 12 weeks
  Individual declares "No" to smoking any form of tobacco product since being discharged from hospital
Self-report of having a smoke-free home at 4 weeks post discharge | 4 weeks
  Individual declares "No" to anyone ever smoking inside home (even by the door or window) at 4 weeks post-discharge
Acceptance and utilization of the different components of enhance intervention | 12 weeks
  Individual declares to have used the different components of the enhanced intervention (has not ticked "didn't use") and declared them to be "1 Very helpful" or "2"
Reduction in number of cigarettes smoked per day at four weeks post-discharge compared to before hospital admission | 4 weeks
  Reduction in number of self reported cigarettes smoked per day at four weeks post-discharge, compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: John Britton, MD, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham City Hospital, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No